CLINICAL TRIAL: NCT07313189
Title: Effect of Stabilizer Pressure Biofeedback on Neck Dysfunction Post Neck Dissection Surgeries
Brief Title: Stabilizer Pressure Biofeedback on Neck Dysfunction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Hager Hussein Noah abdelsamea Shaheen, Demonstrator at Department of Surgery and Burn - Faculty of Physical Therapy - Cairo University, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2151997
Record Dates: First submitted 2025-12-17; First posted 2025-12-31 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2025-12

CONDITIONS: Head and Neck Cancer
Keywords: Biofeedback; Neck dysfunction; Neck dissection surgeries
MeSH Terms: conditions — Head and Neck Neoplasms

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Stabilizer pressure biofeedback plus traditional physical therapy (Experimental): Stabilizer pressure biofeedback plus traditional physical therapy
  Strength Training Protocol for Deep Cervical Flexors Using Pressure Biofeedback Unit (PBU):
  * The air bag of the pressure biofeedback unit was placed under the occiput. Participants instructed to perform a gentle nodding movement in order to reach five target pressure levels between 22 and 30 mmHg.
  * Each pressure level was held for 10 seconds.
  The training program consisted of:
  * 3 sets per session.
  * 10 repetitions in each set.
  * A rest period of two minutes was given between each set to prevent muscle fatigue .
  * Participants received stabilizer pressure biofeedback training 3 sessions per week for 6 weeks.
  The traditional physical therapy program included range of motion exercises, stretching exercises, and strengthening exercises, three times a week for six weeks
  Interventions: Device: Stabilizer pressure biofeedback plus traditional physical therapy
- Traditional physical therapy (Experimental): Traditional Physical Therapy Program The traditional physical therapy program included range of motion exercises, stretching exercises, and strengthening exercises, three times a week for six weeks
  Interventions: Other: Traditional physical therapy

INTERVENTIONS:
Device: Stabilizer pressure biofeedback plus traditional physical therapy — Stabilizer pressure biofeedback
  Strength Training Protocol for Deep Cervical Flexors Using Pressure Biofeedback Unit (PBU):
  * The air bag of the pressure biofeedback unit was placed under the occiput. Participants instructed to perform a gentle nodding movement in order to reach five target pressure levels between 22 and 30 mmHg.
  * Each pressure level held for 10 seconds.
  The training program will consist of:
  * 3 sets per session.
  * 10 repetitions in each set.
  * A rest period of two minutes was given between each set to prevent muscle fatigue .
  * Participants received stabilizer pressure biofeedback training 3 sessions per week for 6 weeks.
  Traditional physical therapy program The traditional physical therapy program included range of motion exercises, stretching exercises, and strengthening exercises, three times a week for six weeks
  Arms: Stabilizer pressure biofeedback plus traditional physical therapy
Other: Traditional physical therapy — Traditional physical therapy program The traditional physical therapy program included range of motion exercises, stretching exercises, and strengthening exercises, three times a week for six weeks .
  Arms: Traditional physical therapy

SUMMARY:
Fifty patients of both genders with age ranged from 30 - 50 years, suffering from neck dysfunction post neck dissection surgeries participated in this study. The participants were randomly selected from the National Cancer Institute, Cairo, Egypt. They were randomly assigned into two equal groups, 25 patients each (study group and control group).

Group A :( Study Group) In this group of the study, received cranio-cervical flexion training utilizing stabilizer pressure biofeedback in addition to traditional physical therapy program (ROM exercises, stretching and strengthening exercises), 3 times a week for 6 weeks.

Group B :( Control Group) In this group of the study, received traditional physical therapy program (ROM exercises, stretching and strengthening exercises), 3 times a week for 6 weeks.

DETAILED DESCRIPTION:
1-Subjects: Fifty patients of both genders with age ranged from 30 - 50 years, suffering from neck dysfunction post neck dissection surgeries participated in this study. The participants were randomly selected from the National Cancer Institute, Cairo, Egypt. They were randomly assigned into two equal groups, 25 patients each (study group and control group).

Group A :( Study Group) In this group of the study, received cranio-cervical flexion training utilizing stabilizer pressure biofeedback in addition to traditional physical therapy program (ROM exercises, stretching and strengthening exercises), 3 times a week for 6 weeks.

Group B :( Control Group) In this group of the study, received traditional physical therapy program (ROM exercises, stretching and strengthening exercises), 3 times a week for 6 weeks.

2) Equipment:

Therapeutic equipment:

1. Stabilizer pressure biofeedback

   Strength Training Protocol for Deep Cervical Flexors Using Pressure Biofeedback Unit (PBU):
   * The air bag of the pressure biofeedback unit was placed under the occiput. Participants were instructed to perform a gentle nodding movement in order to reach five target pressure levels between 22 and 30 mmHg.
   * Each pressure level was held for 10 seconds.

   The training program consisted of:
   * 3 sets per session.
   * 10 repetitions in each set.
   * A rest period of two minutes was given between each set to prevent muscle fatigue.
   * Participants received stabilizer pressure biofeedback training 3 sessions per week for 6 weeks.
2. Traditional physical therapy program The traditional physical therapy program included range of motion exercises, stretching exercises, and strengthening exercises, three times a week for six weeks

Measurement equipment:

1. Arabic version of neck disability index (NDI):

   The Neck Disability Index (NDI) is a self-reported questionnaire designed to assess the functional impact of neck pain on daily activities. It consists of 10 items covering aspects such as personal care, work, driving, and recreation, with each item scored on a 0-5 scale (0 = no disability, 5 = maximum disability). The total NDI score (ranging from 0 to 50) is calculated by summing the item scores, where higher scores indicate greater disability.
2. Goniometer:

   A goniometer is a medical device used to measure the joint angles of the body, providing an objective assessment of a joint's range of motion (ROM). In this study, a standard, handheld goniometer will be used to measure cervical range of motion (CROM), which includes four primary movements: flexion (bending the neck forward), extension (bending the neck backward), lateral flexion (bending the neck to the side), and rotation (turning the head left or right).
3. Stabilizer pressure biofeedback:

The pressure biofeedback device consists of a meter and a flat pocket pneumatic pump, which transfers the force created by deep cervical muscle contractions to the pressure biofeedback device, which measures the pressure in millimeters of mercury (mmHg). A stabilizer pressure biofeedback device will be used to monitor the constant contractile force of the deep neck muscles.

ELIGIBILITY:
Inclusion Criteria:

* The subject selection was according to the following criteria:

  1. Patients' age ranged between 30-50 years.
  2. Both gender participated in this study.
  3. All patients suffered from neck dysfunction (neck pain, limited ROM and disability) following unilateral neck dissection surgeries.
  4. All patients suffered from moderate to severe pain (VAS score > 4).
  5. All patients undergone modified radical NDS or selective NDS.
  6. All patients began the treatment program 2 weeks post neck dissection surgeries
  7. All patients enrolled to the study had their informed consent.

Exclusion Criteria:

* 1- Neck pain due to other underlying conditions such as:

  * Spinal fracture
  * Osteoporosis
  * Spinal cord compression
  * Congenital postural deformities
  * Inflammatory disorders of the spine
  * Spinal infections
  * Significant neurological disorders
  * Rheumatoid arthritis 2- Malignancy 3- Pregnancy 4- History of cervical spine surgery 5- Epilepsy or any psychological disorders

Ages: 30 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2025-09-10 (Actual); Primary Completion 2025-11-20 (Actual); Study Completion 2025-12-15 (Actual)

PRIMARY OUTCOMES:
Deep cervical flexors strength | Measurements were taken at baseline (pre-treatment) and 6 weeks (post-treatment).
  Strength of DCFs was measured using PBU during the Cranio-Cervical Flexion Test (CCFT).
  * The subject lied in a supine position on a firm plinth. A pressure biofeedback unit was placed under the suboccipital region, and the pressure cuff was inflated to 20 mmHg to support the natural cervical lordosis.
  * The subject then instructed to perform a gentle head-nodding movement, similar to saying "yes," which is known as craniocervical flexion.
  * The subject asked to gradually increase the pressure in increments up to a maximum of 10 mmHg above baseline (i.e., up to 30 mmHg), and hold each pressure level for 10 seconds. The highest pressure level that the subject was able to maintain steadily for 10 seconds was considered the strength level of the deep cervical flexors .
  * Measurements were taken at baseline (pre-treatment) and after 6 weeks (post-treatment).

SECONDARY OUTCOMES:
Cervical range of motion | • Measurements were taken at baseline (pre-treatment) and 6 weeks (post-treatment).
  All the cervical spinal ROM measurements were taken with the subject seated upright on a stable chair by goniometer
Neck pain and disability | • The neck disability index was administered at baseline (pre-treatment) and 6 weeks post-intervention to monitor changes in functional impairment
  • The Arabic version of neck disability index (NDI) was used for assessment of neck pain and disability The Neck Disability Index (NDI) is a self-reported questionnaire designed to assess the functional impact of neck pain on daily activities. It consists of 10 items covering aspects such as personal care, work, driving, and recreation, with each item scored on a 0-5 scale (0 = no disability, 5 = maximum disability). The total NDI score (ranging from 0 to 50) is calculated by summing the item scores, where higher scores indicate greater disability

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Physical Therapy, Giza, Egypt